CLINICAL TRIAL: NCT06041269
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Rosnilimab in Subjects with Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study of Efficacy and Safety of Rosnilimab in Subjects with Moderate to Severe Rheumatoid Arthritis (RENOIR)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AnaptysBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB030-203
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
Keywords: PD-1 Agonist; ANB030; RENOIR; Rosnilimab
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rosnilimab SC Dose 1 (Experimental): This arm will receive treatment SC
  Interventions: Drug: Rosnilimab
- Rosnilimab SC Dose 2 (Experimental): This arm will receive treatment SC
  Interventions: Drug: Rosnilimab
- Rosnilimab SC Dose 3 (Experimental): This arm will receive treatment SC
  Interventions: Drug: Rosnilimab
- Placebo (Placebo Comparator): This arm will receive Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosnilimab — PD-1 agonist antibody
  Other Names: ANB030
  Arms: Rosnilimab SC Dose 1; Rosnilimab SC Dose 2; Rosnilimab SC Dose 3
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
RENOIR Study: This study will evaluate the safety, tolerability, and efficacy of Rosnilimab in subjects with moderate to severe Rheumatoid Arthritis (RA)

DETAILED DESCRIPTION:
This study is a Phase 2 Global, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Rosnilimab in Subjects with Moderate to Severe Rheumatoid Arthritis.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 18 years or older
* A diagnosis of Rheumatoid Arthritis based on ACR/EULAR 2010 classification criteria, for at least 3 months before participating in the trial
* Must be receiving treatment with at least 1, but not more than 2 csDMARDs for at least 3 months and be on stable dosages for at least 8 weeks prior to joining and throughout the trial
* Have had an inadequate response to, or loss of response or intolerance to at least 1 conventional synthetic DMARD (csDMARD), biologic DMARD (bDMARD), or targeted synthetic DMARD (tsDMARD) treatment

Key Exclusion Criteria:

* History of an inflammatory joint disease other than Rheumatoid Arthritis
* Prior exposure to a PD-1 or PD-L1 agonist, antagonist, or modulator
* History of cancer within the last 5 years (except for some skin cancers)
* Any known or suspected condition that would compromise immune status
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-11-29 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Mean change from Baseline in 28-Joint Disease Activity Score based on CRP (DAS28-CRP) at Week 12 | Baseline to Week 12
  The DAS28-CRP is a validated composite assessment that assesses RA disease activity based on tender and swollen joint counts of 28 joints

SECONDARY OUTCOMES:
American College of Rheumatology 20% Improvement Criteria (ACR20) response rate at Week 12 | Baseline to Week 12
American College of Rheumatology 50% and 70% Improvement Criteria (ACR50 and ACR70) response rates at Week 12 | Baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (92):
- United States (36):
  - AnaptysBio Investigative Site 10-132, Flagstaff, Arizona
  - AnaptysBio Investigative Site 10-130, Glendale, Arizona
  - AnaptysBio Investigative Site 10-129, Phoenix, Arizona
  - AnaptysBio Investigative Site 10-131, Tucson, Arizona
  - AnaptysBio Investigative Site 10-105, Covina, California
  - Anaptys Bio Investigative Site 10-119, Rancho Mirage, California
  - AnaptysBio Investigative Site 10-113, San Diego, California
  - AnaptysBio Investigative Site 10-127, San Francisco, California
  - AnaptysBio Investigative Site 10-136, Temecula, California
  - AnaptysBio Investigative Site 10-133, Upland, California
  - AnaptysBio Investigative Site 10-112, Whitter, California
  - AnaptysBio Investigative Site 10-103, Aventura, Florida
  - AnaptysBio Investigative Site 10-141, Avon Park, Florida
  - AnaptysBio Investigative Site 10-118, Boynton Beach, Florida
  - AnaptysBio Investigative Site 10-125, Daytona Beach, Florida
  - AnaptysBio Investigative Site 10-122, Homestead, Florida
  - Anaptys Bio Investigative Site 10-142, Miami, Florida
  - AnaptysBio Investigative Site 10-140, Miami, Florida
  - AnaptysBio Investigative Site 10-102, Miami, Florida
  - AnaptysBio Investigative Site 10-124, Plantation, Florida
  - AnaptysBio Investigative Site 10-139, West Palm Beach, Florida
  - AnaptysBio Investigative Site 10-114, Chicago, Illinois
  - AnaptysBio Investigative Site 10-145, Monroe, Louisiana
  - AnaptysBio Investigative Site 10-143, Brookline, Massachusetts
  - AnaptysBio Investigative Site 10-116, Albuquerque, New Mexico
  - AnaptysBio Investigative Site 10-148, Smithfield, North Carolina
  - AnaptysBio Investigative Site 10-146, Middleburg Heights, Ohio
  - AnaptysBio Investigative Site 10-101, Jackson, Tennessee
  - AnaptysBio Investigative Site 10-120, Allen, Texas
  - AnaptysBio Investigative Site 10-107, Colleyville, Texas
  - AnaptysBio Investigative Site 10-123, Katy, Texas
  - AnaptysBio Investigative Site 10-108, Mesquite, Texas
  - AnaptysBio Investigative Site 10-110, Plano, Texas
  - AnaptysBio Investigative Site 10-106, The Woodlands, Texas
  - AnaptysBio Investigative Site 10-121, Tomball, Texas
  - AnaptysBio Investigative Site 10-117, Beckley, West Virginia
- Belgium (4):
  - AnaptysBio Investigative Site 13-102, Anderlecht, Brussels Capital
  - AnaptysBio Investigative Site 13- 105, Liège, Liège
  - AnaptysBio Investigative Site 13-104, Leuven, Vlaams-Braba
  - AnaptysBio Investigative Site 13-103, Antwerp
- Canada (3):
  - AnaptysBio Investigative Site 11-104, Niagara Falls, Ontario
  - AnaptysBio Investigative Site 11-101, Windsor, Ontario
  - AnaptysBio Investigative Site 11-103, Trois-Rivières, Quebec
- Estonia (3):
  - AnaptysBio Investigative Site 71-102, Tallinn, Estonia
  - AnaptysBio Investigative Site 71-101, Tallinn, Estonia
  - AnaptysBio Investigative Site 71-103, Tartu, Tartu
- France (3):
  - AnaptysBio Investigative Site 16-105, Cahors
  - AnaptysBio Investigative Site 16-101, Montpellier
  - AnaptysBio Investigative Site 16-102, Toulouse
- Georgia (6):
  - AnaptysBio Investigative Site 59-101, Tbilisi
  - AnaptysBio Investigative Site 59-105, Tbilisi
  - AnaptysBio Investigative Site 59-104, Tbilisi
  - AnaptysBio Investigative Site 59-106, Tbilisi
  - AnaptysBio Investigative Site 59-102, Tbilisi
  - AnaptysBio Investigative Site 59-103, Tbilisi
- Germany (4):
  - AnaptysBio Investigative Site 17-103, Berlin
  - AnaptysBio Investigative Site 17-102, Hamburg
  - AnaptysBio Investigative Site 17-107, Hanover
  - AnaptysBio Investigative Site 17-105, Herne
- Hungary (4):
  - AnaptysBio Investigative Site 28-104, Budapest, Budapest
  - AnaptysBio Investigative Site 28-103, Debrecen, Hajdú-Bihar
  - AnaptysBio Investigative Site 28-101, Budapest, Pest County
  - Anaptys Bio Investigative Site 28-106, Budapest
- Italy (6):
  - AnaptysBio Investigative Site 20-106, Milan, Lombardy
  - AnaptysBio Investigative Site 20-101, Pavia, PV
  - AnaptysBio Investigative Site 20-104, Bari
  - AnaptysBio Investigative Site 20-110, Milan
  - AnaptysBio Investigative Site 20-105, Novara
  - AnaptysBio Investigative Site 20-108, Roma
- AnaptysBio Investigative Site73-101, Chisinau, Kishinev, Moldova
- Poland (11):
  - AnaptysBio Investigative Site 30-112, Poznan, Greater Poland Voivodeship
  - AnaptysBio Investigative Site 30-105, Poznan, Greater Poland Voivodeship
  - AnaptysBio Investigative Site 30-101, Poznan, Greater Poland Voivodeship
  - AnaptysBio Investigative Site 30-104, Torun, Kuj-pom
  - AnaptysBio Investigative Site 30-103, Nowa Sól, Lubusz Voivodeship
  - AnaptysBio Investigative Site 30-107, Warsaw, Masovian Voivodeship
  - AnaptysBio Investigative Site 30-106, Opole, Opole Voivodeship
  - AnaptysBio Investigative Site 30-102, Bytom, Woj.Slaskie
  - AnaptysBio Investigative Site 30-111, Bialystok
  - AnaptysBio Investigative Site 30-109, Bydgoszcz
  - AnaptysBio Investigative Site 30-108, Warsaw
- Slovakia (3):
  - AnaptysBio Investigative Site 67-101, Košice, Slovakia
  - AnaptysBio Investigative Site 67-102, Martin
  - AnaptysBio Investigative Site 67-103, Piešťany
- Spain (5):
  - AnaptysBio Investigative Site 24-101, Bilbao, Bizkaia
  - AnaptysBio Investigative Site 24-102, Santiago de Compostela, Coruna
  - AnaptysBio Investigative Site 24-105, Córdoba
  - AnaptysBio Investigative Site 24-104, Santiago de Compostela
  - AnaptysBio Investigative Site 24-103, Santiago de Compostela
- AnaptysBio Investigative Site 34-101, Kyiv, Ukraine
- United Kingdom (2):
  - AnaptysBio Investigative Site 27-101, London
  - AnaptysBio Investigative Site 27-102, Manchester

IPD SHARING:
Plan to Share IPD: Yes